CLINICAL TRIAL: NCT05952999
Title: Examining the Intervention Effectiveness of Hospital at Home for Improving Health Outcomes and Experiences for Patients, Clinicians, and Caregivers
Brief Title: Analysis of the Virtual Acute Care at Home Experience
Acronym: HaH
Status: Enrolling by invitation | Type: Observational
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Colleen J Klein, Education & Research Scientist, Center for Advanced Practice, Principal Investigator, OSF Healthcare System
Other Study IDs: 2015255
Record Dates: First submitted 2023-06-28; First posted 2023-07-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Conditions; Infections; Heart Failure; Renal and Urinary Disorders; Diabetes; Hypertension; Fever; Bronchitis; Asthma, Chronic Obstructive Pulmonary Disease (COPD)
Keywords: home hospital; hospital at home; hospital in the home
MeSH Terms: conditions — Disease; Infections; Heart Failure; Urologic Diseases; Diabetes Mellitus; Hypertension; Fever; Bronchitis; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital at Home Care: The population for this study includes adult patients who are acutely ill and presenting to the emergency room, and are discharged to their home for hospital-level care in the home setting. The patients in this cohort may also include those who are discharged from the hospital early, but receive hospital-level care in the home setting.
  Interventions: Other: Digital Care Solution as supportive personalized care
- Traditional Hospital Care: The population for this study includes adult patients who are acutely ill and presenting to the emergency room who elect not to be discharged, choose to be cared for in the hospital setting.
  Interventions: Other: Traditional Hospital Level Care

INTERVENTIONS:
Other: Digital Care Solution as supportive personalized care — Patients will need to meet screening and inclusion criteria at time of enrollment. As a pragmatic study, researchers will not determine criteria or management of care aspects for patients.
  Other Names: Traditional Hospital Level Care
  Groups: Hospital at Home Care
Other: Traditional Hospital Level Care — Patients will be cared for in the inpatient setting for management of diseases that meet screening and inclusion criteria at time of enrollment for hospital at home. As a pragmatic study, researchers will not determine criteria or management of care aspects for patients.
  Groups: Traditional Hospital Care

SUMMARY:
The purpose of this study is to examine the implementation, intervention effectiveness, and dissemination of a digital acute care delivery model for improving selected health outcomes in the Hospital at Home population.

DETAILED DESCRIPTION:
The investigators will conduct a mixed-methods quasi-experimental research study that will explore the effectiveness of the Hospital at home programs using qualitative interviews and quantitative data as a means to also conduct a process evaluation related to the implementation and efficacy of Hospital at Home programs. The purpose of this pragmatic study is to inform scalability beyond the initial site for implementation within a large healthcare system with a diverse patient population located in various communities, including rural and urban locations.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older who are admitted into the Hospital at Home program after presenting to the emergency department or who are inpatients that can be cared at home for hospital level needs
* Patients meeting the hospital's criteria for admission by diagnosis type (e.g., heart failure, respiratory infections and inflammations, renal failure, diabetes, pneumonia, bronchitis, chronic obstructive pulmonary disease, fever and inflammatory conditions, viral illnesses, other disorders of the nervous system). Diagnoses are determined by clinicians not researchers.
* Patients will need to reside within 30 minutes' drive time from the hospital

Patient caregiver inclusion criteria: (not required for patient participation):

* Age >= 18 years old
* as capacity to consent to study

Clinician or stakeholder inclusion criteria:

* Any member of the home hospital clinical team (a healthcare professional who providing care or equipment for use in the home) who will be participating in delivery of healthcare services,
* Any member of the hospital care teams, including the screening and recruitment of patients for the home hospital intervention and/or providing care to patients that enroll in the intervention that is provided
* Any member of the leadership team who are involved in the operational aspects of program delivery

Exclusion Criteria:

* Need for long-term facility level care or current residence in a facility of this type
* No one will be excluded on the basis of sex or race

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who are receiving care in the hospital at home program and those who are hospitalized but choose to receive hospital care in the home setting after a short period in the hospital. All those enrolled in the Hospital at Home Program will be strategically identified and used as the population for the quantitative and qualitative portions of the study.
Sampling Method: Non-Probability Sample
Enrollment: 9654 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality for patients admitted to digital hospital | Up to 30 days, (date of death from any cause, whichever came first, assessed up to 30 days)
  Total number of deaths over total number of patients admitted to the digital hospital.
30-day readmission rate | Up to 30 days (date of readmission from any cause, whichever came first, assessed up to 30 days)
  Number of 30-day readmissions as defined by Organization using preset criteria
Patient Satisfaction at discharge | up to 1 week
  1-item measure: I would recommend this [insert program name] to others, assessed at discharge name] to others.
Patient Perception of Digital Care at discharge | up to 1 week
  Results of Digital Care - Likert Scale (very satisfied to very dissatisfied)

SECONDARY OUTCOMES:
Escalations (for management and treatment of early decompensation) | up to 2 weeks
  percentage of patients escalated over total hospital digital encounters
Unplanned readmission within 30-days of discharge | up to 30 days
  Number of 30-day readmissions over total number of discharges
Length of Stay | assessed up to 2 weeks
  Day of admission to day of discharge, assessed up to 2 months
Number of participants with Hospital Acquired Infections | assessed up to 1 week
  Number of hospital acquired infections reported (CAUTI, CLABSI, etc.)

OTHER OUTCOMES:
Number of participants with discharge disposition at time of discharge as one other than home | assessed up to 8 weeks
  Exploratory - discharge disposition other than patient's home
Qualitative interviews | through study completion, an average of 2 years
  Interviews with patients, caregivers, and hospital and digital health clinicians, workers, ancillary services
Number of readmissions between discharge and during next 6 months. | Up to 6 months (Re-admission from any cause, assessed up to 6 months)
  Exploratory
Number of Emergency Department visits after discharge for any cause | assessed up to 6 months
  Exploratory
Number of visits in home by provider, clinician, and worker type | assessed up to 2 months
  Exploratory
EuroQol-5D-5L | up to 2 months, assessed twice in this period
  5 items self-reported and visual analogue scale, 0-100, where 100 is the best imaginable health today
Program Implementation and Evaluation Measure | at baseline and 1-year following implementation
  15-item measure to assess health care professionals' perceptions of digital care, measured using a Likert scale of 1 to 5, with 1= Not at all, 2=Slightly, 3=Moderately, 4=Very Much, and 5= Entirely. Includes three open-ended questions
Montgomery caregiver burden inventory measure | at approximately 48 hours following admission and at 31-days post-discharge
  11-items to assess objective, relationship, and stress for caregivers. A 5-point response set ranging from 1 (not at all) to 5 (a great deal)
Clinical Sustainability Assessment Tool | at baseline and 1-year following implementation
  Exploratory - measures organizational and contextual factors for sustainability of a project or initiative. Uses a 7-point Likert scale where 1= to little or no extent to 7=to a great extent. Also includes response option of N/A - not able to answer.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Klein, PhD, APRN, Principal Investigator — OSF HealthCare
Locations (1):
- OSF HealthCare, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arsenault-Lapierre G, Henein M, Gaid D, Le Berre M, Gore G, Vedel I. Hospital-at-Home Interventions vs In-Hospital Stay for Patients With Chronic Disease Who Present to the Emergency Department: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021 Jun 1;4(6):e2111568. doi: 10.1001/jamanetworkopen.2021.11568. PMID 34100939
- [Background] Brody AA, Arbaje AI, DeCherrie LV, Federman AD, Leff B, Siu AL. Starting Up a Hospital at Home Program: Facilitators and Barriers to Implementation. J Am Geriatr Soc. 2019 Mar;67(3):588-595. doi: 10.1111/jgs.15782. Epub 2019 Feb 8. PMID 30735244
- [Background] Chua CMS, Ko SQ, Lai YF, Lim YW, Shorey S. Perceptions of Hospital-at-Home Among Stakeholders: a Meta-synthesis. J Gen Intern Med. 2022 Feb;37(3):637-650. doi: 10.1007/s11606-021-07065-0. Epub 2021 Aug 6. PMID 34363185
- [Background] Cooling M, Klein CJ, Pierce LM, Delinski N, Lotz A, Vozenilek JA. Access to Care: End-to-End Digital Response for COVID-19 Care Delivery. J Nurse Pract. 2022 Feb;18(2):232-235. doi: 10.1016/j.nurpra.2021.09.011. Epub 2021 Sep 25. PMID 34608377
- [Background] Dismore LL, Echevarria C, van Wersch A, Gibson J, Bourke S. What are the positive drivers and potential barriers to implementation of hospital at home selected by low-risk DECAF score in the UK: a qualitative study embedded within a randomised controlled trial. BMJ Open. 2019 Apr 4;9(4):e026609. doi: 10.1136/bmjopen-2018-026609. PMID 30948606
- [Background] Federman AD, Soones T, DeCherrie LV, Leff B, Siu AL. Association of a Bundled Hospital-at-Home and 30-Day Postacute Transitional Care Program With Clinical Outcomes and Patient Experiences. JAMA Intern Med. 2018 Aug 1;178(8):1033-1040. doi: 10.1001/jamainternmed.2018.2562. PMID 29946693
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Savundranayagam MY, Montgomery RJ, Kosloski K. A dimensional analysis of caregiver burden among spouses and adult children. Gerontologist. 2011 Jun;51(3):321-31. doi: 10.1093/geront/gnq102. Epub 2010 Dec 6. PMID 21135026
- [Background] Shelton RC, Chambers DA, Glasgow RE. An Extension of RE-AIM to Enhance Sustainability: Addressing Dynamic Context and Promoting Health Equity Over Time. Front Public Health. 2020 May 12;8:134. doi: 10.3389/fpubh.2020.00134. eCollection 2020. PMID 32478025
- [Background] Yao X, Paulson M, Maniaci MJ, Dunn AN, Nelson CR, Behnken EM, Hart MS, Sangaralingham LR, Inselman SA, Lampman MA, Dunlay SM, Dowdy SC, Habermann EB. Effect of hospital-at-home vs. traditional brick-and-mortar hospital care in acutely ill adults: study protocol for a pragmatic randomized controlled trial. Trials. 2022 Jun 16;23(1):503. doi: 10.1186/s13063-022-06430-6. PMID 35710450
- [Derived] Dalstrom MD, Klein CJ, Rothrock-Magana M, Cooling M. Patient-Centered Care: A Qualitative Analysis of Patient and Caregiver Experiences in a Hospital at Home Program. J Patient Exp. 2025 Jun 2;12:23743735251347706. doi: 10.1177/23743735251347706. eCollection 2025. PMID 40464036